CLINICAL TRIAL: NCT01139060
Title: Organized Self-Management Support Services for Chronic Depression
Acronym: Stride
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kaiser Permanente (Other)
Collaborators: Swedish Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 5R01MH082995 (NIH)
Record Dates: First submitted 2010-06-04; First posted 2010-06-08 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Depression
Keywords: chronic or recurrent depression
MeSH Terms: conditions — Depression; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention Group (Experimental): 18-month organized treatment program focused on outreach and engagement for chronic or recurrent depression
  Interventions: Behavioral: organized care program for chronic or recurrent depression
- Usual Care (No Intervention)

INTERVENTIONS:
Behavioral: organized care program for chronic or recurrent depression
  Arms: Intervention Group

SUMMARY:
The purpose is to test the effectiveness of an organized care program for chronic or recurrent depression. Using a two-arm design, the investigators will randomly assign 300 participants with chronic or recurrent depression to one of two conditions: continued usual care (UC); or an 18-month organized treatment program focused on outreach and engagement, including a weekly group self-management training program, monthly visits with a psychotherapist (in-person or by telephone), and optional one-on-one visits with a peer support specialist. All intervention components are intended as adjuncts to any existing depression treatment (usually antidepressant medication) provided by participants' regular providers.

ELIGIBILITY:
Inclusion Criteria:

* all patients will meet criteria for recurrent major depression or dysthymia

Exclusion Criteria:

* bipolar disorder or psychotic disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 302 (Actual)
Dates: Start 2009-08; Primary Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Evaluate the program's effectiveness, i.e., the effects of the intervention on patient outcomes (depressive symptoms, functional impairment, and disability/lost productivity) and process of care (self-efficacy and self-management behaviors) | 18 months

SECONDARY OUTCOMES:
Examination of moderators of treatment response | 18 months
An estimate of the program's costs and effect on the costs of treatment for depression | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Evette Ludman, PhD, Principal Investigator — Group Health Research Institute
Locations (2):
- United States (2):
  - Group Health Research Insitute, Seattle, Washington
  - Swedish Cherry Hill Clinic, Seattle, Washington

REFERENCES:
- [Derived] Jones SMW, Ludman EJ. Factor Structure and Sensitivity to Change of the Recovery Assessment Scale. J Behav Health Serv Res. 2018 Oct;45(4):690-699. doi: 10.1007/s11414-017-9563-x. PMID 28726086
- [Derived] Ludman EJ, Simon GE, Grothaus LC, Richards JE, Whiteside U, Stewart C. Organized Self-Management Support Services for Chronic Depressive Symptoms: A Randomized Controlled Trial. Psychiatr Serv. 2016 Jan;67(1):29-36. doi: 10.1176/appi.ps.201400295. Epub 2015 Aug 17. PMID 26278222